CLINICAL TRIAL: NCT07035418
Title: Adolescents and Young Adults With Cancer: Their Preferred Involvement in Decision Making
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-58292; NCI-2024-00875 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2025-06-06; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Adolescent Behavior
Keywords: Cancer; Survivor; Adolescent and Young Adults
MeSH Terms: conditions — Adolescent Behavior; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AYA Decision-Making Role Assessment (Experimental): Participants will complete an electronic socio-demographic questionnaire followed by a set of hypothetical clinical decision-making scenarios to assess preferred decision-making roles and involvement of healthcare providers and family/friends. Responses will inform understanding of facilitators and barriers to shared decision-making.
  Interventions: Behavioral: Clinical Decision-Making Scenarios and Preferences Assessment

INTERVENTIONS:
Behavioral: Clinical Decision-Making Scenarios and Preferences Assessment — Participants complete a socio-demographic questionnaire and decision-making preferences scale, including hypothetical clinical scenarios, to identify their preferred decision-making role (active, collaborative, or passive) and the influence of providers or family. Delivered electronically via secure link; reminders sent as needed.

SUMMARY:
The purpose of this mixed-methods study is to determine Adolescent and Young Adult (AYAs) decision making preferences post cancer diagnosis using vignettes designed to assess their preferred involvement in decisions about their cancer treatment and variables associated with these treatment decision-making (TDM) preferences.

ELIGIBILITY:
Inclusion Criteria:

* Age (15-29 years)
* Cancer diagnosis and on therapy, end-of-life or survivors (within 1 year)
* Speaks English
* Reads English
* Cognitively and physically able to participate

Exclusion Criteria:

* Unable to participate in study due to developmental delay or developmental disorder

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Distribution of Decision-Making Roles in Clinical Scenarios | Within 2 weeks of survey link delivery
  Proportion of participants who select an active, collaborative, or passive role in hypothetical clinical decision-making scenarios. Each role will be counted and compared across participant subgroups.

SECONDARY OUTCOMES:
Association Between Sociodemographic Characteristics and Decision-Making Role | At time of electronic survey completion
  This outcome assesses the association between sociodemographic characteristics (e.g., age, race/ethnicity, gender, education level, and employment status) and adolescents' and young adults' preferred treatment decision-making role. Role preference (active, collaborative, or passive) is assessed using the modified Control Preferences Scale. Sociodemographic variables are self-reported via electronic questionnaire. The unit of measure is the chi-square test statistic or ANOVA output, depending on the variable type.
Concordance Between Interview Responses and Scenario-Based Decision-Making Roles | At time of interview, within 4 weeks of survey completion
  Proportion of interview responses that align with or differ from role preferences identified in hypothetical scenarios. Qualitative responses will be coded and categorized into roles for comparison.
Correlation Between Healthcare Encounters and Decision-Making Role Preference | At time of interview, within 4 weeks of survey completion
  This outcome measures the correlation between the number of cancer-related healthcare encounters and adolescents' and young adults' preferred treatment decision-making role. Healthcare encounters will be abstracted from the electronic health record and include clinic visits, procedures, hospitalizations, ICU stays, and emergency department visits. Decision-making role preference (active, collaborative, or passive) will be assessed using the modified Control Preferences Scale. The unit of measure is the Pearson correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Pyke-Grimm, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States